CLINICAL TRIAL: NCT00000531
Title: Antiarrhythmics Versus Implantable Defibrillators (AVID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 74
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2005-05

CONDITIONS: Arrhythmia; Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases; Tachycardia, Ventricular; Ventricular Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Defibrillators, Implantable; Amiodarone; Sotalol

INTERVENTIONS:
Device: defibrillators, implantable
Drug: amiodarone amiodarone
Drug: sotalol

SUMMARY:
To evaluate if use of an implantable cardiac defibrillator (ICD) results in reduction in total mortality, when compared with conventional pharmacological therapy, in patients resuscitated from sudden cardiac death who are otherwise at very high risk of mortality from arrhythmic causes.

DETAILED DESCRIPTION:
BACKGROUND:

Sudden cardiac death is believed to account for a substantial proportion of deaths in patients with evidence of cardiovascular disease. The exact proportion of cardiac deaths that are classified as being sudden varies depending on the population, the underlying disease, and the definition of sudden death. Various estimates suggest that about 500,000 sudden cardiac deaths occur annually in the United States alone. The majority of sudden cardiac deaths are thought to be due to ventricular fibrillation (VF) or tachycardia (VT).

The commonest approach to preventing sudden cardiac death has been by the use of drugs that suppress ventricular ectopy. The rational for this approach is based upon an association between the presence or frequency of ventricular arrhythmia and subsequent mortality in several studies. None of the randomized controlled studies of numerous 'classical' antiarrhythmic agents (other than beta-blockers, which have only a modest effect on arrhythmia suppression) have demonstrated a reduction in sudden or non-sudden cardiac mortality. Indeed, in the recent Cardiac Arrhythmia Suppression Trial (CAST), two class Ic anti-arrhythmic agents demonstrated a 2.5 fold increase in the risk of sudden and non-sudden cardiac deaths despite excellent suppression of ventricular arrhythmia.

Given the disappointing results of most pharmacologic approaches to preventing sudden death, many investigators have turned to non-pharmacologic approaches such as surgery (endocardial resection, stellate ganglionectomy) or the implantation of devices that recognize VT or VF and deliver a shock. The greatest interest has been generated by work on the implantable cardiac defibrillator.

The study was reviewed by an ad hoc working group, the Clinical Applications and Prevention Advisory Committee, and several members of the Cardiology Advisory Committee prior to review and approval by the National Heart, Lung, and Blood Advisory Council in September 1991. The Request for Proposals was released in February 1992.

DESIGN NARRATIVE:

At approximately 28 clinical sites, patients with ventricular tachycardia or ventricular fibrillation were screened. Those with ventricular fibrillation or serious ventricular tachycardia were entered into a registry for long-term mortality follow-up using the National Death Index. Patients with the prospect of long-term benefit from an ICD and/or antiarrhythmic drug therapy and without exclusions to an ICD or to amiodarone and without a transient or correctible cause of the index event were entered into the trial.

Patients meeting the criteria were randomized to treatment with an ICD or treatment with antiarrhythmic drug therapy. Allocation was stratified by clinical site and index arrhythmia, either ventricular fibrillation or ventricular tachycardia. Patients assigned to the antiarrhythmic drug therapy and without contraindications to sotalol underwent subrandomization to either empiric amiodarone or sotalol, the latter treatment guided by either ambulatory monitoring or electrophysiologic testing. Patients who, after subrandomization, had low levels (less than 30 beats per hour) of ventricular ectopic beats and no inducible ventricular arrhythmias at electrophysiologic study were not treated with sotalol and instead received empiric amiodarone. The AVID protocol allowed usual clinical practice but restricted interventions to state-of-the art ICD devices and first-line antiarrhythmic agents to amiodarone and sotalol. Patients who could not take amiodarone were not included in the trial. The protocol encouraged the use of concurrent drugs such as angiotensin-converting enzyme inhibitors, aspirin, and beta-blockers when appropriate, administered before randomization and maintained throughout the study. The primary endpoint was total mortality. Secondary endpoints were cost of health care and quality of life. Nonlethal events such as ICD shock, sustained arrhythmia, or syncope were tabulated.

Patients were followed every three months for assessment of secondary endpoints, to record therapies delivered by the ICD and potential adverse effects of the ICD, and to assess compliance and potential adverse symptoms in patients treated with antiarrhythmic drugs. A 12-lead electrocardiogram was obtained every six months, and appropriate laboratory and pulmonary tests were performed at six and eighteen months on patients receiving amiodarone. The average follow-up was expected to be 2.6 years. Analysis was done by intention-to-treat. The outcome of primary interest in the subrandomization between sotalol and amiodarone was the time to withdrawal from assigned therapy.

After a review of the data by the Data and Safety Monitoring Board, the AVID study was stopped early on April 7, 1997 because of the findings that after one year, patients in the defibrillator group experienced a nearly 38 percent reduction in deaths compared to the group of patients taking an antiarrhythmic drug. The defibrillator group had about a 25 percent reduction in deaths in years two and three.

ELIGIBILITY:
Men & women with VF, VT with syncope, or VT without syncope, but with ejection fraction less than or equal to .40 & systolic blood pressure less than 80 mm Hg, chest pain , or near syncope.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-09; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Hallstrom — University of Washington

REFERENCES:
- [Background] Hallstrom AP, Greene HL, Wyse DG, Zipes D, Epstein AE, Domanski MJ, Schron EB; AVID Investigators. Antiarrhythmics Versus Implantable Defibrillators (AVID)--rationale, design, and methods. Am J Cardiol. 1995 Mar 1;75(7):470-5. PMID 7863991
- [Background] Mower MM. AVID necessity. Pacing Clin Electrophysiol. 1994 Feb;17(2):258-60; author reply 262-6. doi: 10.1111/j.1540-8159.1994.tb01381.x. No abstract available. PMID 7513414
- [Background] Fogoros RN. An AVID dissent. Pacing Clin Electrophysiol. 1994 Nov;17(11 Pt 1):1707-11. doi: 10.1111/j.1540-8159.1994.tb03736.x. PMID 7838777
- [Background] Connolly SJ. "An AVID dissent": commentary. Pacing Clin Electrophysiol. 1994 Nov;17(11 Pt 1):1712-3. doi: 10.1111/j.1540-8159.1994.tb03737.x. PMID 7838778
- [Background] Singer I. AVID necessity. Pacing Clin Electrophysiol. 1994 Feb;17(2):260-2; author reply 262-6. doi: 10.1111/j.1540-8159.1994.tb01382.x. No abstract available. PMID 7513415
- [Background] Brooks MM, Hallstrom A, Peckova M. A simulation study used to design the sequential monitoring plan for a clinical trial. Stat Med. 1995 Oct 30;14(20):2227-37. doi: 10.1002/sim.4780142006. PMID 8552899
- [Background] Curtis AB, Hallstrom AP, Klein RC, Nath S, Pinski SL, Epstein AE, Wyse G, Cannom DS, Renfroe E. Influence of patient characteristics in the selection of patients for defibrillator implantation (the AVID Registry). Antiarrhythmics Versus Implantable Defibrillators. Am J Cardiol. 1997 May 1;79(9):1185-9. doi: 10.1016/s0002-9149(97)00079-9. PMID 9164882
- [Background] Josephson ME, Nisam S. The AVID trial: evidence based or randomized control trials--is the AVID study too late? Antiarrhythmics Versus Implantable Defibrillators. Am J Cardiol. 1997 Jul 15;80(2):194-7. doi: 10.1016/s0002-9149(97)00341-x. PMID 9230158
- [Background] Are implantable cardioverter-defibrillators or drugs more effective in prolonging life? The Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial Executive Committee. Am J Cardiol. 1997 Mar 1;79(5):661-3. No abstract available. PMID 9068527
- [Background] Domanski MJ, Saksena S, Wyse G, Hallstrom A, Schron EB, Nanda A, Nanda A, Kutalek S. Clinical and socioeconomic profile of patients with malignant ventricular arrhythmias in 1993 to 1995. AVID investigators. Antiarrhythmics Versus Implantable Defibrillator. Am J Cardiol. 1997 Aug 1;80(3):299-301. doi: 10.1016/s0002-9149(97)00349-4. PMID 9264422
- [Background] Kim SG, Hallstrom A, Love JC, Rosenberg Y, Powell J, Roth J, Brodsky M, Moore R, Wilkoff B. Comparison of clinical characteristics and frequency of implantable defibrillator use between randomized patients in the Antiarrhythmics Vs Implantable Defibrillators (AVID) trial and nonrandomized registry patients. Am J Cardiol. 1997 Aug 15;80(4):454-7. doi: 10.1016/s0002-9149(97)00394-9. PMID 9285657
- [Background] Antiarrhythmics versus Implantable Defibrillators (AVID) Investigators. A comparison of antiarrhythmic-drug therapy with implantable defibrillators in patients resuscitated from near-fatal ventricular arrhythmias. N Engl J Med. 1997 Nov 27;337(22):1576-83. doi: 10.1056/NEJM199711273372202. PMID 9411221
- [Background] Fogoros RN. Why the antiarrhythmics versus implantable defibrillator (AVID) trial sets the wrong precedent. Am J Cardiol. 1997 Sep 15;80(6):762-5. doi: 10.1016/s0002-9149(97)00510-9. No abstract available. PMID 9315584
- [Background] Jenkins LS, Steinberg JS, Kutalek SP, et al: Quality of life in patients enrolled in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial. Circulation 1997;96:I-439
- [Background] Larsen GC, McAnulty JH, Hallstrom A, et al: Hospitalization charges in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial: the AVID economic analysis study. Circulation 1997;96:I-77
- [Background] Myerburg RJ, Castellanos A. Clinical trials of implantable defibrillators. N Engl J Med. 1997 Nov 27;337(22):1621-3. doi: 10.1056/NEJM199711273372209. No abstract available. PMID 9371860
- [Background] Singer I, Nisam S. There should never be another antiarrhythmics versus implantable defibrillator (AVID) trial. Am J Cardiol. 1997 Sep 15;80(6):766-8. doi: 10.1016/s0002-9149(97)00511-0. No abstract available. PMID 9315585
- [Background] Kimm SG, Love J, Rosenberg Y, Powell J, AVID Investigators: Therapy in the AVID (Antiarrhythmics Versus Implantable Defibrillators) Trial is not signifcantly different from current clinical practice. Circulation 1995;92:I782
- [Background] Brooks MM, Jenkins LS, Schron EB, Steinberg JS, Cross JA, Paeth DS. Quality of life at baseline: is assessment after randomization valid? The AVID Investigators. The Antiarrhythmics Versus Implantable Defibrillators. Med Care. 1998 Oct;36(10):1515-9. doi: 10.1097/00005650-199810000-00009. PMID 9794344
- [Background] Anderson JL, Hallstrom AP, Epstein AE, Pinski SL, Rosenberg Y, Nora MO, Chilson D, Cannom DS, Moore R. Design and results of the antiarrhythmics vs implantable defibrillators (AVID) registry. The AVID Investigators. Circulation. 1999 Apr 6;99(13):1692-9. doi: 10.1161/01.cir.99.13.1692. PMID 10190878
- [Background] Domanski MJ, Sakseena S, Epstein AE, Hallstrom AP, Brodsky MA, Kim S, Lancaster S, Schron E. Relative effectiveness of the implantable cardioverter-defibrillator and antiarrhythmic drugs in patients with varying degrees of left ventricular dysfunction who have survived malignant ventricular arrhythmias. AVID Investigators. Antiarrhythmics Versus Implantable Defibrillators. J Am Coll Cardiol. 1999 Oct;34(4):1090-5. doi: 10.1016/s0735-1097(99)00327-7. PMID 10520795
- [Background] Epstein AE, Powell J, Yao Q, Ocampo C, Lancaster S, Rosenberg Y, Cannom DS, Herre JM, Greene HL. In-hospital versus out-of-hospital presentation of life-threatening ventricular arrhythmias predicts survival: results from the AVID Registry. Antiarrhythmics Versus Implantable Defibrillators. J Am Coll Cardiol. 1999 Oct;34(4):1111-6. doi: 10.1016/s0735-1097(99)00305-8. PMID 10520799
- [Background] Causes of death in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial. J Am Coll Cardiol. 1999 Nov 1;34(5):1552-9. doi: 10.1016/s0735-1097(99)00376-9. PMID 10551706
- [Background] Exner DV, Reiffel JA, Epstein AE, Ledingham R, Reiter MJ, Yao Q, Duff HJ, Follmann D, Schron E, Greene HL, Carlson MD, Brodsky MA, Akiyama T, Baessler C, Anderson JL. Beta-blocker use and survival in patients with ventricular fibrillation or symptomatic ventricular tachycardia: the Antiarrhythmics Versus Implantable Defibrillators (AVID) trial. J Am Coll Cardiol. 1999 Aug;34(2):325-33. doi: 10.1016/s0735-1097(99)00234-x. PMID 10440140
- [Background] Pinski SL, Yao Q, Epstein AE, Lancaster S, Greene HL, Pacifico A, Cook JR, Jadonath R, Marinchak RA. Determinants of outcome in patients with sustained ventricular tachyarrhythmias: the antiarrhythmics versus implantable defibrillators (AVID) study registry. Am Heart J. 2000 May;139(5):804-13. doi: 10.1016/s0002-8703(00)90011-5. PMID 10783213
- [Background] Raitt MH, Renfroe EG, Epstein AE, McAnulty JH, Mounsey P, Steinberg JS, Lancaster SE, Jadonath RL, Hallstrom AP; Antiarrhythmics Versus Implantable Defibrillators investigators. "Stable" ventricular tachycardia is not a benign rhythm : insights from the antiarrhythmics versus implantable defibrillators (AVID) registry. Circulation. 2001 Jan 16;103(2):244-52. doi: 10.1161/01.cir.103.2.244. PMID 11208684
- [Background] Kron J, Herre J, Renfroe EG, Rizo-Patron C, Raitt M, Halperin B, Gold M, Goldner B, Wathen M, Wilkoff B, Olarte A, Yao Q. Lead- and device-related complications in the antiarrhythmics versus implantable defibrillators trial. Am Heart J. 2001 Jan;141(1):92-8. doi: 10.1067/mhj.2001.111261. PMID 11136492
- [Background] Exner DV, Sheldon RS, Pinski SL, Kron J, Hallstrom A. Do baseline characteristics accurately discriminate between patients likely versus unlikely to benefit from implantable defibrillator therapy? Evaluation of the Canadian implantable defibrillator study implantable cardioverter defibrillatory efficacy score in the antiarrhythmics versus implantable defibrillators trial. Am Heart J. 2001 Jan;141(1):99-104. doi: 10.1067/mhj.2001.111768. PMID 11136493
- [Background] Hallstrom AP, McAnulty JH, Wilkoff BL, Follmann D, Raitt MH, Carlson MD, Gillis AM, Shih HT, Powell JL, Duff H, Halperin BD; Antiarrhythmics Versus Implantable Defibrillator (AVID) Trial Investigators. Patients at lower risk of arrhythmia recurrence: a subgroup in whom implantable defibrillators may not offer benefit. Antiarrhythmics Versus Implantable Defibrillator (AVID) Trial Investigators. J Am Coll Cardiol. 2001 Mar 15;37(4):1093-9. doi: 10.1016/s0735-1097(00)01208-0. PMID 11263614
- [Background] Epstein AE. AVID necessity. Pacing Clin Electrophysiol. 1993 Sep;16(9):1773-5. doi: 10.1111/j.1540-8159.1993.tb01808.x. No abstract available. PMID 7692406
- [Background] Hallstrom AP, Anderson JL, Cobb LA, Friedman PL, Herre JM, Klein RC, McAnulty J, Steinberg JS. Advantages and disadvantages of trial designs: a review of analysis methods for ICD studies. AVID Investigators. Pacing Clin Electrophysiol. 2000 Jun;23(6):1029-38. doi: 10.1111/j.1540-8159.2000.tb00892.x. PMID 10879390
- [Background] Exner DV, Pinski SL, Wyse DG, Renfroe EG, Follmann D, Gold M, Beckman KJ, Coromilas J, Lancaster S, Hallstrom AP; AVID Investigators. Antiarrhythmics Versus Implantable Defibrillators. Electrical storm presages nonsudden death: the antiarrhythmics versus implantable defibrillators (AVID) trial. Circulation. 2001 Apr 24;103(16):2066-71. doi: 10.1161/01.cir.103.16.2066. PMID 11319196
- [Background] Hickey K, Curtis AB, Lancaster S, Larsen G, Warwick D, McAnulty J, Mitchell LB. Baseline factors predicting early resumption of driving after life-threatening arrhythmias in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial. Am Heart J. 2001 Jul;142(1):99-104. doi: 10.1067/mhj.2001.115787. PMID 11431664
- [Background] Akiyama T, Powell JL, Mitchell LB, Ehlert FA, Baessler C; Antiarrhythmics versus Implantable Defibrillators Investigators. Resumption of driving after life-threatening ventricular tachyarrhythmia. N Engl J Med. 2001 Aug 9;345(6):391-7. doi: 10.1056/NEJM200108093450601. PMID 11496849
- [Background] Smith TW. Driving after ventricular arrhythmias. N Engl J Med. 2001 Aug 9;345(6):451-2. doi: 10.1056/NEJM200108093450609. No abstract available. PMID 11496857
- [Background] Wyse DG, Love JC, Yao Q, Carlson MD, Cassidy P, Greene LH, Martins JB, Ocampo C, Raitt MH, Schron E, Stamato NJ, Olarte A. Atrial fibrillation: a risk factor for increased mortality--an AVID registry analysis. J Interv Card Electrophysiol. 2001 Sep;5(3):267-73. doi: 10.1023/a:1011460631369. PMID 11500581
- [Background] Steinberg JS, Martins J, Sadanandan S, Goldner B, Menchavez E, Domanski M, Russo A, Tullo N, Hallstrom A; AVID Investigators. Antiarrhythmic drug use in the implantable defibrillator arm of the Antiarrhythmics Versus Implantable Defibrillators (AVID) Study. Am Heart J. 2001 Sep;142(3):520-9. doi: 10.1067/mhj.2001.117129. PMID 11526368
- [Background] Beumont PJ, Richards DH, Gelder MG. A study of minor psychiatric and physical symptoms during the menstrual cycle. Br J Psychiatry. 1975 May;126:431-4. doi: 10.1192/bjp.126.5.431. No abstract available. PMID 1168516
- [Background] Wyse DG, Friedman PL, Brodsky MA, Beckman KJ, Carlson MD, Curtis AB, Hallstrom AP, Raitt MH, Wilkoff BL, Greene HL; AVID Investigators. Life-threatening ventricular arrhythmias due to transient or correctable causes: high risk for death in follow-up. J Am Coll Cardiol. 2001 Nov 15;38(6):1718-24. doi: 10.1016/s0735-1097(01)01597-2. PMID 11704386
- [Background] Schron EB, Exner DV, Yao Q, Jenkins LS, Steinberg JS, Cook JR, Kutalek SP, Friedman PL, Bubien RS, Page RL, Powell J. Quality of life in the antiarrhythmics versus implantable defibrillators trial: impact of therapy and influence of adverse symptoms and defibrillator shocks. Circulation. 2002 Feb 5;105(5):589-94. doi: 10.1161/hc0502.103330. PMID 11827924
- [Background] Larsen G, Hallstrom A, McAnulty J, Pinski S, Olarte A, Sullivan S, Brodsky M, Powell J, Marchant C, Jennings C, Akiyama T; AVID Investigators. Cost-effectiveness of the implantable cardioverter-defibrillator versus antiarrhythmic drugs in survivors of serious ventricular tachyarrhythmias: results of the Antiarrhythmics Versus Implantable Defibrillators (AVID) economic analysis substudy. Circulation. 2002 Apr 30;105(17):2049-57. doi: 10.1161/01.cir.0000015504.57641.d0. PMID 11980684
- [Background] Cook JR, Rizo-Patron C, Curtis AB, Gillis AM, Bigger JT Jr, Kutalek SP, Coromilas J, Hofer BI, Powell J, Hallstrom AP; AVD Investigators. Effect of surgical revascularization in patients with coronary artery disease and ventricular tachycardia or fibrillation in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Registry. Am Heart J. 2002 May;143(5):821-6. doi: 10.1067/mhj.2002.121732. PMID 12040343
- [Background] Renfroe EG, Heywood G, Foreman L, Schron E, Powell J, Baessler C, Warwick D, Morris M, Hallstrom A; AVID Coordinators and Investigators. Antiarrhythmics Versus Implantable Defibrillators. The end-of-study patient survey: methods influencing response rate in the AVID Trial. Control Clin Trials. 2002 Oct;23(5):521-33. doi: 10.1016/s0197-2456(02)00225-8. PMID 12392866
- [Background] Raitt MH, Klein RC, Wyse DG, Wilkoff BL, Beckman K, Epstein AE, Coromilas J, Friedman PL, Martins J, Ledingham RB, Greene HL; Antiarrhythmics Versus Implantable Defibrillators Investigators. Comparison of arrhythmia recurrence in patients presenting with ventricular fibrillation versus ventricular tachycardia in the Antiarrhythmics Versus Implantable Defibrillators (AVID) trial. Am J Cardiol. 2003 Apr 1;91(7):812-6. doi: 10.1016/s0002-9149(03)00015-8. PMID 12667566
- [Background] Brodsky MA, Mitchell LB, Halperin BD, Raitt MH, Hallstrom AP; AVID Investigators. Prognostic value of baseline electrophysiology studies in patients with sustained ventricular tachyarrhythmia: the Antiarrhythmics Versus Implantable Defibrillators (AVID) trial. Am Heart J. 2002 Sep;144(3):478-84. doi: 10.1067/mhj.2002.125502. PMID 12228785
- [Background] Steinberg JS, Beckman K, Greene HL, Marinchak R, Klein RC, Greer SG, Ehlert F, Foster P, Menchavez E, Raitt M, Wathen MS, Morris M, Hallstrom A. Follow-up of patients with unexplained syncope and inducible ventricular tachyarrhythmias: analysis of the AVID registry and an AVID substudy. Antiarrhythmics Versus Implantable Defibrillators. J Cardiovasc Electrophysiol. 2001 Sep;12(9):996-1001. doi: 10.1046/j.1540-8167.2001.00996.x. PMID 11573709
- [Background] Hallstrom A, Friedman L, Denes P, Rizo-Patron C, Morris M; CAST Investigators; AVID Investigators. Do arrhythmia patients improve survival by participating in randomized clinical trials? Observations from the Cardiac Arrhythmia Suppression Trial (CAST)and the Antiarrhythmics Versus Implantable Defibrillators Trial (AVID). Control Clin Trials. 2003 Jun;24(3):341-52. doi: 10.1016/s0197-2456(03)00002-3. PMID 12757998
- [Background] Mitchell LB, Powell JL, Gillis AM, Kehl V, Hallstrom AP; AVID Investigators. Are lipid-lowering drugs also antiarrhythmic drugs? An analysis of the Antiarrhythmics versus Implantable Defibrillators (AVID) trial. J Am Coll Cardiol. 2003 Jul 2;42(1):81-7. doi: 10.1016/s0735-1097(03)00498-4. PMID 12849664
- [Background] Klein RC, Schron EB, Renfroe EG, Hallstrom A, Kron J, Ocampo C, Leonen A, Tullo N; Avid Investigators. Factors determining ICD implantation in drug therapy patients after termination of antiarrythmics versus implantable defibrillators trial. Pacing Clin Electrophysiol. 2003 Dec;26(12):2235-40. doi: 10.1111/j.1540-8159.2003.00353.x. PMID 14675006
- [Background] Klein RC, Raitt MH, Wilkoff BL, Beckman KJ, Coromilas J, Wyse DG, Friedman PL, Martins JB, Epstein AE, Hallstrom AP, Ledingham RB, Belco KM, Greene HL; AVID Investigators. Analysis of implantable cardioverter defibrillator therapy in the Antiarrhythmics Versus Implantable Defibrillators (AVID) Trial. J Cardiovasc Electrophysiol. 2003 Sep;14(9):940-8. doi: 10.1046/j.1540-8167.2003.01554.x. PMID 12950538
- [Background] Page RL, Zipes DP, Powell JL, Luceri RM, Gold MR, Peters R, Russo AM, Bigger JT Jr, Sung RJ, McBurnie MA; AVID Investigators. Seasonal variation of mortality in the Antiarrhythmics Versus Implantable Defibrillators (AVID) study registry. Heart Rhythm. 2004 Oct;1(4):435-40. doi: 10.1016/j.hrthm.2004.06.001. PMID 15851196
- [Background] Zipes DP. Implantable cardioverter-defibrillator. Lifesaver or a device looking for a disease? Circulation. 1994 Jun;89(6):2934-6. doi: 10.1161/01.cir.89.6.2934. No abstract available. PMID 8205712
- Available data/document: Individual Participant Data Set: AVID — http://biolincc.nhlbi.nih.gov/studies/avid/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/avid/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/avid/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/avid/